CLINICAL TRIAL: NCT04553133
Title: PHASE 1/2A DOSE ESCALATION, FINDING AND EXPANSION STUDY EVALUATING SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS AND ANTI TUMOR ACTIVITY OF PF-07104091 AS A SINGLE AGENT AND IN COMBINATION THERAPY
Brief Title: PF-07104091 as a Single Agent and in Combination Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4161001; 2024-515492-34-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-08-21; First posted 2020-09-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Small Cell Lung Cancer; Ovarian Cancer; Breast Cancer
Keywords: Hormone receptor-positive human epidermal growth factor receptor 2 negative breast cancer; Cyclin-Dependent Kinase 2 Inhibitor; PF-07104091; palbociclib; letrozole; cyclin-dependent kinase; Ibrance
MeSH Terms: conditions — Small Cell Lung Carcinoma; Ovarian Neoplasms; Breast Neoplasms | interventions — palbociclib; Fulvestrant; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- PF-07104091 (Experimental): CDK2 monotherapy dose escalation
  Interventions: Drug: PF-07104091 monotherapy dose escalation
- PF-07104091 + palbociclib + fulvestrant (Experimental): CDK2 + palbociclib + fulvestrant
  Interventions: Drug: PF-07104091 + palbociclib + fulvestrant
- PF-07104091 + palbociclib + letrozole (Experimental): CDK2 + palbociclib + letrozole
  Interventions: Drug: PF-07104091 + palbociclib + letrozole
- PF-07104091 monotherapy dose expansion (SCLC) (Experimental): PF-07104091 monotherapy dose expansion (SCLC)
  Interventions: Drug: PF-07104091 monotherapy dose expansion (SCLC)
- PF-07104091 monotherapy dose expansion (ovarian) (Experimental): PF-07104091 monotherapy dose expansion (ovarian)
  Interventions: Drug: PF-07104091 monotherapy dose expansion (ovarian)
- PF-07104091 + fulvestrant (post CDK4/6) dose expansion (Experimental): PF-07104091 + fulvestrant (post CDK4/6) dose expansion
  Interventions: Drug: PF-0704091 + Fulvestrant (post CDK4/6)
- PF-07104091 + fulvestrant (post CDK 4/6) dose escalation (Experimental): CDK2+ fulvestrant (post CDK 4/6) dose escalation
  Interventions: Drug: PF-07104091 + Fulvestrant (post CDK4/6)

INTERVENTIONS:
Drug: PF-07104091 monotherapy dose escalation — PF-07104091 will be administered orally
  Arms: PF-07104091
Drug: PF-07104091 + palbociclib + fulvestrant — PF-07104091 will be administered orally in combination with palbociclib and fulvestrant
  Arms: PF-07104091 + palbociclib + fulvestrant
Drug: PF-07104091 + palbociclib + letrozole — PF-07104091 will be administered orally in combination with palbociclib and letrozole
  Arms: PF-07104091 + palbociclib + letrozole
Drug: PF-07104091 monotherapy dose expansion (ovarian) — PF-07104091 will be administered orally
  Arms: PF-07104091 monotherapy dose expansion (ovarian)
Drug: PF-07104091 monotherapy dose expansion (SCLC) — PF-07104091 will be administered orally
  Arms: PF-07104091 monotherapy dose expansion (SCLC)
Drug: PF-07104091 + Fulvestrant (post CDK4/6) — PF-07104091 will be administered orally in combination with fulvestrant
  Arms: PF-07104091 + fulvestrant (post CDK 4/6) dose escalation
Drug: PF-0704091 + Fulvestrant (post CDK4/6) — PF-07104091 + fulvestrant (post 4/6) dose expansion
  Arms: PF-07104091 + fulvestrant (post CDK4/6) dose expansion

SUMMARY:
To assess the safety and tolerability of increasing doses of PF-07104091 and to estimate the Maximum Tolerated Dose (MTD) and/or select the Recommended Phase 2 dose (RP2D) for PF-07104091 as a single agent in participants with advanced or metastatic small cell lung, breast and ovarian cancers.

DETAILED DESCRIPTION:
Study C4161001 is a Phase 1, open label, multi dose, multi center, dose escalation, safety, pharmacokinetic (PK) and pharmacodynamic study of PF-07104091 in adult patients with advanced or metastatic small cell lung cancer (SCLC), advanced platinum resistant epithelial ovarian cancer/fallopian tube cancer/primary peritoneal cancer, locally recurrent/advanced or metastatic triple negative breast cancer (TNBC), HR-positive HER2-negative advanced or mBC, advanced or metastatic non-small cell lung cancer (NSCLC). This two part study will assess the safety and tolerability of increasing dose levels of PF-07104091 in Part 1, and establish the recommended Phase 2 dose (RP2D) in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Participants with HR-positive HER2-negative advanced or metastatic breast cancer (received at least two prior lines in the advanced or metastatic setting including one prior line of combined CDK4/6 inhibitor and endocrine therapy and no more than two prior lines of cytotoxic chemotherapy)
* Participants with locally recurrent/advanced or metastatic TNBC who have received up to 2 prior lines of chemotherapy in the advanced or metastatic setting
* Participants with advanced platinum resistant epithelial ovarian cancer (EOC)/fallopian tube cancer/primary peritoneal cancer (PPC) (histologically or cytologically proven) who have received at least 1 systemic anti-cancer therapy containing a platinum analog
* Participants with cytological diagnosis of advanced/metastatic SCLC
* Participants with or cytological diagnosis of advanced/metastatic NSCLC
* Participants with HR-positive HER2-negative advanced or metastatic breast cancer (second line plus setting) (histologically or cytologically proven).
* Participants entering the study in the expansion cohort have at least one measurable lesion as defined by RECIST version 1.1 that has not been previously irradiated
* Performance Status 0 or 1
* Adequate bone marrow, hematological, kidney and liver function
* Resolved acute effects of any prior therapy to baseline severity

Exclusion Criteria:

* Participants with known symptomatic brain metastases requiring steroids
* Participants with any other active malignancy within 3 years prior to enrollment
* Major surgery within 3 weeks prior to study entry
* Radiation therapy within 3 weeks prior to study entry.
* Systemic anti cancer therapy within 4 weeks prior to study
* Prior irradiation to >25% of the bone marrow
* Participants with active, uncontrolled bacterial, fungal, or viral infection, including HBV, HCV, and known HIV or AIDS related illness
* Active COVID-19/SARS-CoV2 infection
* Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
* Any of the following in the previous 6 months: myocardial infarction, long QT syndrome, Torsade de Pointes, arrhythmias, serious conduction system abnormalities, unstable angina, coronary/peripheral artery bypass graft, symptomatic CHF, New York Heart Association class III or IV, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism, and/or other clinical significant episode of thrombo embolic disease.
* Anticoagulation with vitamin K antagonists or factor Xa inhibitors is not allowed.
* Hypertension that cannot be controlled by medications
* Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry.
* Known or suspected hypersensitivity to active ingredient/excipients in PF 07104091.
* Active inflammatory gastrointestinal disease, chronic diarrhea, known diverticular disease or previous gastric resection or lap band surgery.
* Participants with advanced/metastatic, symptomatic, visceral spread, that are at risk of life threatening complications in the short
* Participants with an indwelling catheter that has an external component such as those used for drainage of effusion(s) or central venous catheter that is externally
* Previous high dose chemotherapy requiring stem cell rescue
* Known abnormalities in coagulation such as bleeding diathesis, or treatment with anticoagulants precluding intramuscular injections of goserelin (if applicable).
* Current use or anticipated need for food or drugs that are known strong CYP3A4/5 or UGT1A9 inhibitors or inducers
* Current use or anticipated need for drugs that are known sensitive UGT1A1 substrates with narrow therapeutic
* Serum pregnancy test positive at screening
* Other medical or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Number of participants with Dose-limiting toxicities (DLT) during first cycle | 28 days
  Number of participants with DLTs, which are typically Grade 3 or higher adverse events will be summarized by dose level
To evaluate incidence of treatment emergent adverse events and laboratory abnormalities | From baseline until end of study treatment or study completion (approximately 2 years)
  Type, incidence, severity, timing, seriousness and relationship to study treatment of adverse events and any laboratory abnormalities will be summarized by dose level
Evaluate pulse rate that is out of normal range and changes in pulse rate as compared to baseline | From baseline until end of study treatment or study completion (approximately 2 years)
  Identify pulse rate readings that are outside the normal range. The number and percentage of participants who experienced significant pulse rate change from baseline will be summarized by dose level
Evaluate blood pressure that is out of normal range and changes in blood pressure as compared to baseline | From baseline until end of study treatment or study completion (approximately 2 years)
  Identify systolic and diastolic readings that are outside the normal range. The number and percentage of participants who experienced significant blood pressure change from baseline will be summarized by dose level
To evaluate heart rate corrected QT interval and changes in corrected QT interval as compared to baseline | From baseline until end of study treatment or study completion (approximately 2 years)
  Determine the effect of the drug on QT prolongation. The number and percentage of participants who experienced QT interval prolongation will be summarized by dose level
To evaluate the preliminary antitumor activity of PF-07104091 as a single agent and in combination with palbociclib and in combination with letrozole or fulvestrant or fulvestrant alone by objective response rate (ORR) in dose expansion | From baseline through disease progression or study completion (approximately 2 years)
  Percentage of participants with a best overall response of complete response (CR) or partial response (PR) using RECIST 1.1

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of PF-07104091 after a single dose and multiple dose | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
  Peak concentration of PF-07104091 during selected cycles
Time to maximum plasma concentration (Tmax) of PF-07104091 after a single dose and multiple dose | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
  Time to peak concentration of PF-07104091 during selected cycles
Area under the concentration versus time curve from time zero to the last quantifiable time point prior to the next dose (AUClast) of PF-07104091 | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
  AUC of PF-07104091 will be calculated at selected cycles
Area under the curve of PF-07104091 with or without food | From baseline through time to event on study or study completion (approximately 2 years)
  AUC of PF-07104091 in plasma and whether absorption of the drug is affected when taken by food
Maximum plasma concentration of PF-07104091 with or without food | From baseline through time to event on study or study completion (approximately 2 years)
  Peak concentrations of PF-07104091 in plasma and whether absorption of the drug is affected when taken by food
To document any preliminary evidence of antitumor activity of PF-07104091 as a single agent and in combination with palbociclib and in combination with letrozole or fulvestrant or fulvestrant alone by objective response rate (ORR) in dose escalation | From baseline and every 8 weeks through disease progression or study completion (approximately 2 years)
  Percentage of participants with a best overall response of CR or PR using RECIST 1.1
To document any preliminary evidence of antitumor activity of PF-07104091 by time to event endpoints | From baseline through time to event on study or study completion (approximately 2 years)
  Time from first assessment of event endpoint to last assessment of using RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (33):
  - Medical Oncology & Hematology Associates DBA Mission Cancer and Blood, Clive, Iowa
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - Medical Oncology & Hematology Associates DBA Mission Cancer and Blood, Des Moines, Iowa
  - Norton Cancer Institute Downtown, Louisville, Kentucky
  - Norton Cancer Institute Pharmacy, Downtown Pharmacy, Louisville, Kentucky
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Norton Cancer Institute, St. Matthews, Louisville, Kentucky
  - Norton Women's and Children's Hospital (St. Matthews), Louisville, Kentucky
  - Norton Cancer Institute, Audubon, Louisville, Kentucky
  - Norton Hospital (Audubon), Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Brownsboro Campus, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center (IDS Pharmacy), Long Island City, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura & Isaac Perlmutter Cancer Center - NYU ACC, New York, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - MSK Rockefeller Outpatient Pavilion, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - White Plains Hospital, White Plains, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - UVA Breast Care Center, Charlottesville, Virginia
- Argentina (3):
  - Centro Oncologico Korben, Caba, Buenos Aires
  - Fundación Cenit Para La Investigación En Neurociencias, CABA, Buenos Aires F.D.
  - Centro Polivalente de Asistencia e Investigacion Clinica - CER San Juan, San Juan
- Bulgaria (3):
  - Specialized Hospital for Active Treatment of Oncology - Haskovo, Haskovo
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Complex Oncology Center - Shumen, Shumen
- China (4):
  - Jilin Province Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4161001